CLINICAL TRIAL: NCT06976177
Title: A Multi-center, Open, Single-arm Phase IIb Clinical Study to Evaluate the Safety and Efficacy of MT1013 Injection for the Treatment of Secondary Hyperparathyroidism (SHPT) Patients With Chronic Kidney Disease Undergoing Maintenance Dialysis
Brief Title: Study of MT1013 Injection for the Treatment of Secondary Hyperparathyroidism (SHPT) Patients With Chronic Kidney Disease Undergoing Maintenance Dialysis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT1013-II-C02
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Secondary Hyperparathyroidism (SHPT) in Subjects With Chronic Kidney Disease (CKD) on Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MT1013 (Experimental): MT1013 injection administered intravenously (IV) three times per week for 52(Part A) or 26(Part B) weeks
  Interventions: Drug: MT1013

INTERVENTIONS:
Drug: MT1013 — MT1013 is a novel calcimimetic agent

SUMMARY:
This is a multi-center, open, single-arm phase IIb clinical study comprising 2 parts, which Part A will enroll about 110 subjects, and Part B will enroll about 190 subjects to investigate long-term efficacy and safety of MT1013 after treatment.The treatment duration for Part A MAD study is 52 weeks and the duration for Part B study is 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject capable of understanding written information ,willing to participate in, and provide a written informed consent; 2.Male or female subjects must be at least 18 years old when signing the informed consent; 3.The subjects must undergo maintenance hemodialysis three times a week or five times two weeks for at least three months； 4.Dialysate calcium concentration≥1.25 mmol/L (2.5 mEq/L); 5.Diagnosed of Secondary Hyperparathyroidism (SHPT);

Exclusion Criteria:

* 1.Primary hyperparathyroidism; 2.Refusal to discontinue cinacalcet, etelcalcetide, or other calcimimetics during the study; 3.Has used RANKL inhibitors such as denosumab within 6 months before screening. 4.Diagnosed with gastrointestinal bleeding within 6 months prior to screening; 5.Subjects with severe uncontrolled hypertension, defined as systolic blood pressure>180 mmHg and/or diastolic blood pressure>110 mmHg, despite optimal drug treatment prior to enrollment; 6.The subjects underwent parathyroidectomy within 6 months prior to screening, or plan to undergo parathyroidectomy during the study; 7.Subjects are allergic or intolerant to any component of the investigational drug； 8.History of epileptic seizures or ongoing epilepsy related treatment within 1 year prior to screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-08-19 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
The occurrence of adverse events within 26 weeks | Baseline up to 26 weeks
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

SECONDARY OUTCOMES:
Percentage of participants with iPTH during 150-300pg/mL at week 26 | at week 26

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China